CLINICAL TRIAL: NCT01519050
Title: Predictors of Postoperative Left Ventricular Function in Patients Undergoing Mitral Valve Repair for Severe Degenerative Mitral Regurgitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: KEK ZH 2011- 0274
Record Dates: First submitted 2012-01-23; First posted 2012-01-26 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Severe Degenerative Mitral Regurgitation
MeSH Terms: interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: mitral valve repair — Mitral valve repair in patients with degenerative mitral regurgitation

SUMMARY:
The aim of the study is to investigate whether a predictive score (combination of several validated predictors) better predicts postoperative left ventricular function than any single predictor in patients undergoing mitral valve repair for degenerative mitral regurgitation.

A single center, prospective cohort study

ELIGIBILITY:
Inclusion criteria:

* Age 18- 85 years
* Patients with severe degenerative mitral regurgitation undergoing mitral valve repair at our institution

Exclusion criteria:

* Functional or ischemic mitral regurgitation
* Presence of relevant (symptomatic) Coronary Artery Disease
* Inability of exercising on semi supine bicycle

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients with mitral valve proplapse ondergoing mitral valve repair for severe mitral regurgitation
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Patric Biaggi, MD, Senior physican, Principal Investigator — University Hospital Zurich, Division of Cardiology
Locations (1):
- University Hospital Zurich, Division of Cardiology, Zurich, Canton of Zurich, Switzerland